CLINICAL TRIAL: NCT00000852
Title: A Pilot Study of Allogeneic Lymphocyte Transfer in HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: DATRI 016
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: T-Lymphocytes; Acquired Immunodeficiency Syndrome; Transplantation, Homologous; Immunotherapy, Adoptive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Procedure: Allogeneic lymphocyte transfer

SUMMARY:
To examine, in HIV-infected patients, the safety of allogeneic lymphocyte transfer (i.e., infusion of white blood cells taken from an HIV-negative parent, sibling, or adult offspring who has a compatible blood type). To measure the distribution and survival of allogeneic lymphocytes in the circulation of HIV-infected patients, and to determine whether their infusion results in enhanced immunity. To determine whether enhanced immunity is passively transferred or actively induced.

There is evidence that periodic infusion of allogeneic lymphocytes obtained from the peripheral blood of HLA-matched HIV-1 seronegative siblings of patients with AIDS can, in some instances, restore the number of circulating CD4+ lymphocytes. However, more controlled studies are needed to better quantitate the immunologic reconstitution seen with this type of therapy.

DETAILED DESCRIPTION:
There is evidence that periodic infusion of allogeneic lymphocytes obtained from the peripheral blood of HLA-matched HIV-1 seronegative siblings of patients with AIDS can, in some instances, restore the number of circulating CD4+ lymphocytes. However, more controlled studies are needed to better quantitate the immunologic reconstitution seen with this type of therapy.

Lymphocytes obtained by leukapheresis from a healthy, HIV-negative parent, sibling, or adult offspring of the HIV-infected patient are infused at day 0 and at weeks 4 and 8. A small portion of the lymphocytes obtained at day 0 will be radiolabeled prior to infusion, and two total body scans will be performed. Patients also undergo two tonsillar biopsies. Patients are followed weekly for 16 weeks, then by telephone periodically for 3 years (at 1 year, 2 years, 2.5 years, and 3 years).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Stable antiretroviral therapy.

Allowed:

* Maintenance therapy for a controlled opportunistic infection.

Patients must have:

* HIV infection.
* CD4 count 50-200 cells/mm3.
* No ongoing major opportunistic infections.
* Been on stable antiretroviral therapy for the past 2 months.
* Tonsils present.
* Life expectancy greater than 6 months.
* An HLA-single haplotype matched, single haplotype mismatched parent, sibling, or adult offspring who is ABO, Rh compatible to serve as an HIV-negative lymphocyte donor.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Lymphoma or other malignancy requiring chemotherapy.
* Bleeding disorder that would preclude a tonsillar biopsy.
* Antibody on donor/recipient lymphocyte reactive antibody assay.

Donors with the following symptoms or conditions are excluded:

* Medical condition that would endanger health of donor or recipient.
* Failure to meet established donor standards on blood screening tests.
* CMV seropositivity if the patient (recipient) is CMV seronegative.
* Pregnancy.

Concurrent Medication:

Excluded:

* GM-CSF or G-CSF.
* Any investigational drug.
* Immunomodulators (such as interferon, steroids, topical corticosteroids, thalidomide, pentoxifylline, IL-2).
* Nonsteroidal anti-inflammatory drugs.
* Aspirin.

Prior Treatment:

Excluded:

* Blood transfusion within the past 2 months.

Required:

* Stable antiretroviral therapy for at least 2 months prior to study entry.

Active substance abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12

CONTACTS AND LOCATIONS:
Overall Officials: Lederman M, Study Chair; Lee E, Study Chair; Deyton L, Study Chair
Locations (1):
- Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio, United States

REFERENCES:
- [Background] Volunteers sought for HIV treatment study. NIAID AIDS Agenda. 1996 Sep:3. PMID 11363923